CLINICAL TRIAL: NCT04994054
Title: Effect of Silkworms (Bombyx Mori L.) Pupae Extracts on Musculoskeletal Biomarkers in Adults With With Relatively Low Muscle Mass: a Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Effect of Silkworms (Bombyx Mori L.) Pupae Extracts on Musculoskeletal Biomarkers in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2021-023
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- silkworms (Bombyx mori L.) pupae extracts group (Experimental): This group takes silkworms (Bombyx mori L.) pupae extracts for 12 weeks.
  Interventions: Dietary Supplement: silkworms (Bombyx mori L.) pupae extracts group
- Placebo group (Placebo Comparator): This group takes placebo for 12 weeks.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: silkworms (Bombyx mori L.) pupae extracts group — silkworms (Bombyx mori L.) pupae extracts 2,400 mg/day for 12 weeks
  Arms: silkworms (Bombyx mori L.) pupae extracts group
Dietary Supplement: Placebo group — Placebo 2,400 mg/day for 12 weeks
  Arms: Placebo group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of silkworms (Bombyx mori L.) pupae extracts on muscle strength, muscle mass, and muscle function in adults with relative sarcopenia for 12 weeks.

DETAILED DESCRIPTION:
A previous study has indicated that silkworms (Bombyx mori L.) pupae extracts may increase muscle mass and strength. Therefore, the investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of silkworms (Bombyx mori L.) pupae extracts on muscle strength, muscle mass, and muscle function in adults with relative sarcopenia; the safety of the compound are also evaluated. The Investigators examine the peak torque/body weight at 60°/s knee extension, handgrip strength, skeletal muscle mass, physical performance, and metabolic parameters at baseline, as well as after 12 weeks of intervention. Fifty four adults were administered either 2,400 mg of silkworms (Bombyx mori L.) pupae extracts or a placebo each day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* <110% of the standard lean body mass as measured using the body composition analyzer
* Body mass index (BMI) ranging from 18.5 to 30.0 kg/m2

Exclusion Criteria:

* Vegetarian
* History of any central bone fracture within 1 year
* History of cancer or serious cerebro-cardiovascular diseases within 6 months
* Abnormal liver or renal function (more than twice the normal upper limit of the research institute)
* Uncontrolled diabetes mellitus (>160 mg/dL of fasting blood sugar)
* Uncontrolled hypertension (>160/100 mmHg)
* Uncontrolled thyroid diseases.
* History of medication for psychiatric diseases such as severe affective disorder, schizophrenia, and substance use.
* Alcohol abuser
* Allergic reaction to constituent foods
* Severe gastrointestinal symptoms such as heartburn and indigestion
* Those who are pregnant, lactating, or planning to become pregnant during the clinical trial
* Those who have participated in other drug clinical trials within the last 3months

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
the peak torque at 60°/s knee extension (/kg) | 12 weeks
  conducted on the Biodex System 3 Pro isokinetic dynamometer (Biodex, Inc.)

SECONDARY OUTCOMES:
appendicular skeletal mass/(height x height) | 12 weeks
  using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
appendicular skeletal mass/weight x 100 | 12 weeks
  using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
skeletal Muscle Mass Index/(height x height) | 12 weeks
  using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
concentration of creatinine kinase (IU/L) | 12 weeks
  creatinine kinase (IU/L) measured at baseline and after 12 weeks
concentration of creatine (mg/dL) | 12 weeks
  creatine (mg/dL) measured at baseline and after 12 weeks
EuroQol five dimensional five levels | 12 weeks
  an index of life quality, minimum, maximum values (-0.171, 1), higher scores mean a better outcome, which will be measured at baseline and after 12 weeks
handgrip strength (kg), right and left | 12 weeks
  using a hydraulic hand dynamometer (Jamar)
body weight (kg) | 12 weeks
  using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
skeletal musle mass (kg) | 12 weeks
  using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
total fat percent (%) | 12 weeks
  using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks
truncal fat percent (%) | 12 weeks
  using dual-energy X-ray absorptiometry measured at baseline and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi JI, Kweon HY, Lee YL, Lee JH, Lee SY. Efficacy of Silkworm Pupae Extract on Muscle Strength and Mass in Middle-Aged and Older Individuals: A Randomized, Double-Blind, Placebo-Controlled Trial. J Nutr Health Aging. 2023;27(7):578-585. doi: 10.1007/s12603-023-1942-9. PMID 37498105